CLINICAL TRIAL: NCT02375841
Title: Coping With Glioblastoma: A Study of Communication Between Physicians, Patients, and Caregivers
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-034
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Brain Cancer; Glioblastoma
Keywords: Communication; Physicians; Patients; Caregivers; 15-034
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Communication | interventions — Psychometrics; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Physicians, Patients, and Caregivers: This is a longitudinal study of patients with GBM with recurrent or multi-recurrent disease as determined by their neuro-oncologist (on the basis of clinical and/or radiological findings). Patients will indicate a single caregiver who will consent separately and perform separate assessments. The study assessments will evaluate the content of the discussion in which this change in disease status was communicated, as well as include patient-reported and caregiver-reported outcomes. We intend to accrue 160 total participants (80 patients and 80 caregivers) with complete post-discussion visit follow-ups over 18-24 months.
  Interventions: Behavioral: psychometric tests, questionnaires and neurocognitive assessments

INTERVENTIONS:
Behavioral: psychometric tests, questionnaires and neurocognitive assessments

SUMMARY:
The purpose of this study is to learn more about the way physicians communicate with brain tumor patients. This study will look at how oncologists provide information about brain tumors, brain scan results, and treatment options. This study will look at how oncologists provide information about brain tumors, brain scan results, and treatment options. Ultimately, the investigators hope to use these findings to improve communication between patients, caregivers and their doctors.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria:

* 18 years or older
* Pathologic diagnosis of WHO grade IV glioma, as per MSKCC medical record or outside medical record.
* In the judgment of the consenting professional, proficiency in English that will allow the participant to be able to complete study questionnaires and assessments. Many of the study assessments are available only in English.
* At the time of consent, orientation to self, place, month and year

Caregiver Inclusion Criteria:

* 18 years or older
* Identified by the patient as a relative, friend, or partner with whom he or she has a significant relationship and who provides him or her informal (unpaid) care (i.e., physical or emotional assistance).
* In the judgment of the consenting professional, proficiency in English that will allow to complete study questionnaires and assessments. Many of the study assessments are available only in English.

Oncologist Inclusion Criteria:

* Treating Neuro-Oncologist in the Department of Neurology

Exclusion Criteria:

Patient Exclusion Criteria:

* A patient will be excluded if in the opinion of his/her attending neuro-oncologist or the covering neuro-oncologist, he does not have the capacity to consent to the study based on clinical evaluation
* Aphasia precluding comprehension and verbalization of consent to participate, in the estimation of the attending physician.

Caregiver Exclusion Criteria:

* There are no caregiver exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with GBM will be screened in the outpatient clinic at MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
number of responses from patients, to 3 yes/no questions | 2 years
  The curability of the patient's cancer (curability) The patient's prognosis (prognosis)The patient's goals of care should his/her condition worsen and he/she becomes critically ill (EOL)
number of responses from caregivers to 3 yes/no questions | 2 years
  The curability of the patient's cancer (curability) The patient's prognosis (prognosis)The patient's goals of care should his/her condition worsen and he/she becomes critically ill (EOL)
number of responses from physicians to 3 yes/no questions | 2 years
  The curability of the patient's cancer (curability) The patient's prognosis (prognosis)The patient's goals of care should his/her condition worsen and he/she becomes critically ill (EOL)

CONTACTS AND LOCATIONS:
Overall Officials: Eli Diamond, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Vermont Medical Center, Burlington, Vermont

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/